CLINICAL TRIAL: NCT05550870
Title: Effect of Raw Versus Roasted Fenugreek Seed Powder in Reducing Blood Glucose Levels in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Sanaullah Iqbal, Associate Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Raw versus Roasted Fenugreek
Record Dates: First submitted 2022-06-20; First posted 2022-09-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
Keywords: Fenugreek; Diabetes; HbA1c; Hyperglycemia; Blood glucose; Raw versus Roasted fenugreek; Type 2 Diabetes; Lipid profile; Cholesterol; Triglycerides; HDL; LDL
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: There are two groups, Group 1 will be given raw fenugreek and group 2 will be given roasted fenugreek. Results will be compared to baselines.
Who Masked: Participant
Masking Description: It is a single-blind clinical trial, in which patients know that fenugreek is being given to them but which form either raw or roasted is unknown to them
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will be given Raw Fenugreek seed powder. The dose will be 7.5grams two times a day i.e, before breakfast and before dinner for the period of three months.
  Interventions: Dietary Supplement: Raw fenugreek seed powder
- Group 2 (Experimental): Group 2 will be given Roasted Fenugreek seed powder, 7.5 grams twice a day before breakfast and dinner for the period of three months.Total number of arms will be 2.
  Interventions: Dietary Supplement: Roasted fenugreek seed powder

INTERVENTIONS:
Dietary Supplement: Raw fenugreek seed powder — It will be given to group 1
  Arms: Group 1
Dietary Supplement: Roasted fenugreek seed powder — It will be given to group 2
  Arms: Group 2

SUMMARY:
Diabetes is a metabolic disorder that causes high glucose levels in the blood and leads to various complications with time such as Retinopathy, neuropathy, and nephropathy, and puts a lot of burden on the health of a person as well as economy of country. Fenugreek is being used for decades in the treatment of various diseases and disorders including diabetes. With the advancement of medical nutrition therapy and processing techniques, it is being used in roasted or cooked form. But previous studies indicate that processing like roasting decrease the fiber content of fenugreek seed and this fiber mainly galactomannan is responsible for reducing hyperglycemia. Another study tells us that in raw form the glycemic index is lowered as compared to roasted or other forms.According to another study the antioxidant activity is increased in roasted form as compared form. So in this study, a clinical trial will be done on two groups of 15 type 2 diabetic patients each that have neither other complications nor on insulin therapy. These total 30 patients Height, Weight, BMI, Fasting and Random Blood sugars, HbA1c, and lipid profile will be checked before the study and after 3 months of a clinical trial. Group 1 will be given Raw fenugreek seed powder and group 2 will be given Roasted fenugreek seed powder 7.5 grams twice a day.The study will be single blinded.

DETAILED DESCRIPTION:
Diabetes mellitus is a metabolic disorder that is marked by high glucose levels in the blood because of insulin resistance or inability of the pancreas to make enough insulin for proper working of carbohydrate metabolism. It is easily obvious from the literature that its prevalence is increasing day by day and in future it seems to rise more. Its complications lead to more problematic situation for the health of diabetic person itself and the economy with each day. Its management includes diet, physical activity and medications. As a dietary component different spices are being used for years like cinnamon and fenugreek. Many people use fenugreek in various forms like its incorporation in chapatti, Indian dish Dosa and others but the form of fenugreek is still un known based on the effectiveness that either it will be more beneficial in cooked form like roasting or in raw form for reducing hyperglycemia, because many people take it in roasted form as it decreases its bitterness. As fenugreek is cheap it is of major concern of many diabetic patients for diabetes management.

This study is aimed to determine the effect of Raw versus Roasted Fenugreek seed powder in reducing the blood glucose levels in Type 2 Diabetic patients which will be evidenced by Fasting Blood Glucose, Random Blood Glucose and HbA1c

OBJECTIVE of the study is:

1. To explore the potential of Raw and Roasted fenugreek against biomarkers of Type 2 Diabetes in Diabetic Patients.

The methodology of the study comprises of three different phases. Phase 1: Processing of fenugreek Phase 2: Assessment of diabetic patients regards to inclusion and exclusion criteria and groups assignment along with fenugreek sachets Phase 3: Assessment of biochemical tests and anthropometric measurements at the end of the study

Phase 1: Processing of fenugreek Fenugreek will be brought form the local market and will be cleaned for the stones and straws. Fenugreek seeds will be roasted in oven at approximately 130 ± 5 °C for 7 minutes with stirring at regular intervals with laddle so that it will properly and uniformly roasted and it will turn to slight brownish colour along with peculiar aroma. Raw and Roasted fenugreek seeds will be grounded in grinder to get uniform sized flour. Flours will be collected and stored in air tight food grade containers separately for further use at ambient temperature.

Phase 2: Assessment of diabetic patients regards to inclusion and exclusion criteria and groups assignment along with fenugreek sachets

Subjects:

For the study the diabetic patients will be gathered in the diabetic camp at Lahore where their anthropometric and blood sample collection will be done. The participants will be divided in to two groups Group 1 and group 2 with equal participants of 15 in each group. Total 30 patients of Type 2 Diabetes will be selected for this clinical trial .The inclusion criteria include age ranging from 30-50 years old male and female type 2 diabetic patients from Lahore with informed consent and Patients with Diabetes diagnosed from past 5- 15 years. The exclusion criteria consist of: Anyone suffering from any other chronic disease like Cardiac, Pulmonary and Chronic Renal Disease and patients other than inclusion criteria, any diabetic patients on Insulin therapy and Pregnant and Breastfeeding women. Any one suffering from chickpeas, peanut or coriander allergy. Height, weight and BMI of all patients will be checked as anthropometric measures. Patients BMI will be classified according to WHO criteria.

Whereas BMI =Weight in kg/Height in meter squares. Random, fasting blood sugars will be tested along with HbA1c and Lipid profile. The participants will be divided in to two groups one with Raw fenugreek and second with Roasted one. The duration of the study will be 3 months.

Experimental design:

Group 1 will be given Raw Fenugreek in Ziploc sachets of 7.5 grams (2 sachets for a day equals to 15 grams) for every 2 weeks, ultimately for period of 3 months. Bimonthly their Fasting and Random Blood sugar will be checked also. Participants will be told to take 1 sachet before breakfast and one before dinner. Similarly Group 2 will be given the Roasted fenugreek in the same manner as that of group 1.The participants will be allowed to take their regular oral medications like metformin for diabetes. There will be a gap of 1-2 hours between oral medications (oral hypoglycemic agents) and fenugreek intake as its fiber becomes mucilaginous and can interfere with the drug activity.

Biochemical testing:

Anthropometric measurements such as height weight and BMI will be checked at baseline, and after three months. Besides the anthropometry, the study participant's Fasting and Random Blood glucose levels will be checked before, after every two weeks and after completion of the study. In addition after every 2 weeks through Glucometer by using finger prick method. Before, and at the end of the study HbA1c will be checked also. Patients Blood Lipid Profile will also be checked before and after the study.

Phase 3: Assessment of biochemical tests and anthropometric measurements at the end of the study At the end of the study, HbA1c along with fasting and Random Blood Sugars will be tested so that effectiveness of both groups to their baselines can be compared after the study. Lipid profile will also be monitored and compared to the base lines. Their height, weight and BMI will also be monitored at the end of the study and will be compared to the baselines.

Statistical analysis:

Statistical Package for Social Science software (version 22) will be used for the analysis of data. Independent t test will be applied to check the differences between group 1 and group 2 at baseline. Paired t test will be used to check the differences between baselines and final results after treatment within a group. One way ANOVA will also be used.The level of significance will be <0.05

ELIGIBILITY:
Inclusion Criteria:

- 30-50 years of Type 2 Diabetic patients with past 5-15 years of diabetes Type 2

Exclusion Criteria:

* Any patient on insulin therapy
* Patients with other chronic diseases like Cardiac, Renal, or Pulmonary diseases.
* Pregnant and Lactating mothers
* Anyone with peanut or coriander allergy or Allergy to Fabeace Family

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Expected change in the level of HbA1c . | 3 months
  HbA1c will be assessed after three months of trial through a blood sample
Weight will be checked in kg | 3 months
  weight machine will be used to assess weight in both groups after 3 months
BMI will be checked in kg/^2 | 3 months
  BMI after study will be assessed as kg/m2
Fasting Blood Sugar in mg/dl | Bimonthly till 3 months
  After every two weeks the fasting blood sugar will be assessed via Glucometer
Random Blood Sugar in mg/dl | Bimonthly till 3 months
  Bimonthly Random blood sugar will be assessed via Glucometer
HDL in mg/dl | 3 months
  High Density Lipoprotein-Cholesterol will be assessed after the study in a private lab
LDL in mg/dl | 3 months
  Low Density Lipoprotein-Cholesterol will be tested after the intervention period
Triglycerides in mg/dl | 3 months
  Triglycerides will be tested after the intervention period
Cholesterol in mg/dl | 3 months
  Cholesterol will be tested after the intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- University of Veterinary and Animal Sciences, Paksitan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelwahab NS, Morsi A, Ahmed YM, Hassan HM, AboulMagd AM. Ecological HPLC method for analyzing an antidiabetic drug in real rat plasma samples and studying the effects of concurrently administered fenugreek extract on its pharmacokinetics. RSC Adv. 2021 Jan 25;11(8):4740-4750. doi: 10.1039/d0ra08836f. eCollection 2021 Jan 21. PMID 35424379
- [Background] Ahmad A, Amir RM, Ameer K, Ali SW, Siddique F, Hayat I, Ahmad Z, Faiz F. 2020. Ameliorative effects of fenugreek (Trigonella foenum-graecum) seed on type 2 diabetes. Food Sci. Technol.(AHEAD).
- [Background] Ahmad H, Kashif S, Afreen A, Safdar M, Ahmed Z. 2021. Comparative effect of Fenugreek and Cinnamon on management of newly diagnosed cases of Type-2 Diabetes Mellitus. Food Sci. Technol.
- [Background] Alshali KZ. 2020. Review of herb supplement use in type 2 diabetes. Archives of Pharmacy Practice. 11(2).
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S62-9. doi: 10.2337/dc10-S062. No abstract available. PMID 20042775
- [Background] Ansari R, Ansari S. 2011. Effectiveness of fenugreek for lowering hemoglobin (HbA1c) in patients with self-management of type 2 diabetes: a randomized, controlled trial. Medical Complications of Type. 2: 393-412.
- [Background] Baset ME, Ali TI, Elshamy H, El Sadek AM, Sami DG, Badawy MT, Abou-Zekry SS, Heiba HH, Saadeldin MK, Abdellatif A. 2020. Anti-diabetic effects of fenugreek (Trigonella foenum-graecum): A comparison between oral and intraperitoneal administration - an animal study. Int J Funct Nutr. 1(1): 2.
- [Background] Chatterjee S, Khunti K, Davies MJ. Type 2 diabetes. Lancet. 2017 Jun 3;389(10085):2239-2251. doi: 10.1016/S0140-6736(17)30058-2. Epub 2017 Feb 10. PMID 28190580
- [Background] Das S, Dhananjaya BL, Desiraju S. 2018. Trigonella foenum-graceum (fenugreek) for Management of Diabetes. Int. j. biochem. res. 14(3): 1-10.
- [Background] Gupta RC, Chang D, Nammi S, Bensoussan A, Bilinski K, Roufogalis BD. Interactions between antidiabetic drugs and herbs: an overview of mechanisms of action and clinical implications. Diabetol Metab Syndr. 2017 Jul 26;9:59. doi: 10.1186/s13098-017-0254-9. eCollection 2017. PMID 28770011
- [Background] Haber SL, Keonavong J. Fenugreek use in patients with diabetes mellitus. Am J Health Syst Pharm. 2013 Jul 15;70(14):1196, 1198, 1200, 1202-3. doi: 10.2146/ajhp120523. No abstract available. PMID 23820455
- [Background] Hassani SS, Fallahi Arezodar F, Esmaeili SS, Gholami-Fesharaki M. Effect of Fenugreek Use on Fasting Blood Glucose, Glycosylated Hemoglobin, Body Mass Index, Waist Circumference, Blood Pressure and Quality of Life in Patients with Type 2 Diabetes Mellitus: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trials. Galen Med J. 2019 Mar 30;8:e1432. doi: 10.31661/gmj.v8i0.1432. eCollection 2019. PMID 34466512
- [Background] Jiang JX, Zhu LW, Zhang WM, Sun RC. 2007. Characterization of Galactomannan Gum from Fenugreek (Trigonella foenum-graecum) Seeds and Its Rheological Properties. Int. J. Polym. 56(12): 1145-1154.
- [Background] Kharroubi AT, Darwish HM. Diabetes mellitus: The epidemic of the century. World J Diabetes. 2015 Jun 25;6(6):850-67. doi: 10.4239/wjd.v6.i6.850. PMID 26131326
- [Background] Khursheed R, Singh SK, Wadhwa S, Kapoor B, Gulati M, Kumar R, Ramanunny AK, Awasthi A, Dua K. Treatment strategies against diabetes: Success so far and challenges ahead. Eur J Pharmacol. 2019 Nov 5;862:172625. doi: 10.1016/j.ejphar.2019.172625. Epub 2019 Aug 23. PMID 31449807
- [Background] Kumar K, Kumar S, Datta A, Bandyopadhyay A. 2015. Effect of fenugreek seeds on glycemia and dyslipidemia in patients with type 2 diabetes mellitus. Int. j. health med. 4(7): 997-1000.
- [Background] Majeed M, Majeed S, Nagabhushanam K, Arumugam S, Natarajan S, Beede K, Ali F. Galactomannan from Trigonella foenum-graecum L. seed: Prebiotic application and its fermentation by the probiotic Bacillus coagulans strain MTCC 5856. Food Sci Nutr. 2018 Feb 20;6(3):666-673. doi: 10.1002/fsn3.606. eCollection 2018 May. PMID 29876118
- [Background] Pandey H, Awasthi P. Effect of processing techniques on nutritional composition and antioxidant activity of fenugreek (Trigonella foenum-graecum) seed flour. J Food Sci Technol. 2015 Feb;52(2):1054-60. doi: 10.1007/s13197-013-1057-0. Epub 2013 Jun 12. PMID 25694718
- [Background] Pradeep SR, Srinivasan K. Amelioration of hyperglycemia and associated metabolic abnormalities by a combination of fenugreek (Trigonella foenum-graecum) seeds and onion (Allium cepa) in experimental diabetes. J Basic Clin Physiol Pharmacol. 2017 Sep 26;28(5):493-505. doi: 10.1515/jbcpp-2015-0140. PMID 28599386
- [Background] Ranade M, Mudgalkar N. A simple dietary addition of fenugreek seed leads to the reduction in blood glucose levels: A parallel group, randomized single-blind trial. Ayu. 2017 Jan-Jun;38(1-2):24-27. doi: 10.4103/ayu.AYU_209_15. PMID 29861588
- [Background] Sanlier N, Gencer F. 2020. Role of spices in the treatment of diabetes mellitus: A minireview. Trends Food Sci Technol . 99: 441-449.
- [Background] Sarwar S, Hanif MA, Ayub MA, Boakye YD, Agyare C. 2020. Fenugreek. In. Medicinal Plants of South Asia. Elsevier. p. 257-271.
- [Background] Sharma R. 1986. Effect of fenugreek seeds and leaves on blood glucose and serum insulin responses in human subjects. Nutr Res 6(12): 1353-1364.
- [Background] Srinivasan K. 2019. Chapter 3.15 - Fenugreek (Trigonella foenum-graecum L.) Seeds Used as Functional Food Supplements to Derive Diverse Health Benefits. In: Nabavi SM, Silva AS, editors. Nonvitamin and Nonmineral Nutritional Supplements. Academic Press. p. 217-221.
- [Background] Standl E, Khunti K, Hansen TB, Schnell O. The global epidemics of diabetes in the 21st century: Current situation and perspectives. Eur J Prev Cardiol. 2019 Dec;26(2_suppl):7-14. doi: 10.1177/2047487319881021. PMID 31766915
- [Background] Suchitra M, Parthasarathy S. 2015. Effect of administration of fenugreek seeds on HbA1C levels in uncontrolled diabetes mellitus-a randomized controlled trial. Int J Pharm Tech Res. 8(2): 180-182.